CLINICAL TRIAL: NCT00180999
Title: Randomised Study to Compare the Effect of r-Hu-EPO Administration With Transfusion of Red Blood Cell Concentrates and Also With the Administration of Polyvitamins in Anemic and Tired Patients Presenting a Bad Prognostic in Middle Course
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUMFATIGUE; CSET 98/663
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: - Medico-Economic Aspects (Evaluation of Medical Costs Related to the Three Strategies and Evaluation of Cost/Efficacy)

INTERVENTIONS:
Drug: Erythropoiétine

SUMMARY:
Randomised study to compare the effect of r-Hu-EPO administration with transfusion of Red Blood cell concentrates and also with the administration of polyvitamins in anemic and tired patients presenting a bad prognostic in middle course.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* 18-70 yrs
* metastatic or locally advanced cancer
* Life expectancy > 3 months
* hemoglobin between 7 and 10 g/100ml
* no contraindication to r-Hu-EPO
* with written informed consent at entry time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420
Dates: Start 2002-02

PRIMARY OUTCOMES:
Quality of life, in particular when related to tiredness (FACT F)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie LAPIERRE, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave-Roussy, Villejuif, France